CLINICAL TRIAL: NCT04493372
Title: Deciphering Preserved Autonomic Function After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan J. Solinsky, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-005772
Record Dates: First submitted 2020-07-17; First posted 2020-07-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; Autonomic Imbalance; Autonomic Dysreflexia; Orthostatic Hypotension
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Hypotension, Orthostatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individuals with spinal cord injury (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of sympathetic activation; Diagnostic Test: Testing of autonomic dysreflexia
- Individuals without spinal cord injury (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of sympathetic activation; Diagnostic Test: Testing of autonomic dysreflexia

INTERVENTIONS:
Diagnostic Test: Tests of sympathetic inhibition — Bolus phenylephrine infusion using the Oxford technique will generate the need to inhibit sympathetic activity. Similarly, resting state Mayer waves will be assessed with regard to heart rate and blood pressure responses.
Diagnostic Test: Tests of sympathetic activation — Cold pressor test of the hand will be used to cause sympathetic activation. Valsalva's maneuver will assess the ability to buffer against blood pressure fall (phase II).
Diagnostic Test: Testing of autonomic dysreflexia — Cold pressor test of the foot and bladder pressor response (in individuals with SCI) will be tested.

SUMMARY:
This study looks to characterize gradients of dysfunction in the autonomic nervous system after spinal cord injury. The autonomic nervous system plays key roles in regulation of blood pressure, skin blood flow, and bladder health- all issues that individuals with spinal cord injury typically suffer. Focusing on blood pressure regulation, the most precise metric with broad clinical applicability, the investigators will perform laboratory-based tests to probe the body's ability to generate autonomic responses. For both individuals with spinal cord injury and uninjured controls, laboratory-based experiments will utilize multiple parallel recordings to identify how the autonomic nervous system is able to inhibit and activate signals. The investigators anticipate that those with autonomic dysfunction after spinal cord injury will exhibit abnormalities in these precise metrics. The investigators will further have research participants wear a smart watch that tracks skin electrical conductance, heart rate, and skin temperature, which can all provide clues as to the degree of autonomic dysfunction someone may suffer at home. The investigators will look to see if any substantial connections exist between different degrees of preserved autonomic function and secondary autonomic complications from spinal cord injury. In accomplishing this, the investigators hope to give scientists important insights to how the autonomic nervous system works after spinal cord injury and give physicians better tools to manage these secondary autonomic complications.

DETAILED DESCRIPTION:
This study looks to characterize gradients of dysfunction in the autonomic nervous system after spinal cord injury. To accomplish this, we are enrolling both individuals with and without spinal cord injuries (see inclusion criteria). Individuals will undergo the listed diagnostics as part of a battery of laboratory testing. These will be correlated to clinical histories of autonomic dysfunction the ADFSCI and COMPASS-31 surveys (noted in outcome measures).

ELIGIBILITY:
Inclusion Criteria:

All subjects

- age 18-50 years old.

Participants with spinal cord injury

* Adult onset, traumatic spinal cord injury.
* American Spinal Injury Association Impairment Scale, A-D, to encompass a spectrum of autonomic dysfunction after spinal cord injury.
* Neurological level of injury, C1-T12, as defined by the International Standards for Neurological Classification of Spinal Cord Injury. Incorporating level of injury down to T12 to encompass a broad range of autonomic dysfunction.

Exclusion Criteria:

* History of cardiovascular disease, hypertension, neurologic disorders (with exception of spinal cord injury), or diabetes.
* Women who are pregnant or lactating.
* Currently taking blood thinners.
* Pacemaker, implanted defibrillator, or intrathecal pump incompatible with MRI scanning.
* Cognitive issues preventing informed consent for participation.
* Body mass index >30 kg/m2 for controls, in an effort to limit effects of early cardiovascular disease and diabetes in control population. Body mass index has not proven to be a good estimate of these factors following spinal cord injury.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Valsalva Maneuver Phase II | During laboratory diagnostic testing session
  Presence or absence of phase II on Valsalva maneuver testing, which takes approximately 15 seconds to complete. This will be repeated x3.

SECONDARY OUTCOMES:
Beat-to-beat heart rate | During laboratory diagnostic testing session
  Electrocardiogram will record continuous measures with changes in R-R interval (ms) quantified and compared to baseline.
Beat-to-beat blood pressure | During laboratory diagnostic testing session
  Non-invasive continuous blood pressure monitors will be used, with changes in systolic and diastolic pressure (in mmHg) from resting baseline measured.
Continuous galvanic skin response | During laboratory diagnostic testing session
  Changes from resting state conductance with be quantified with a smartwatch.
Continuous wrist temperature | During laboratory diagnostic testing session
  Changes from resting state temperature with be quantified with a smartwatch.
Quantify autonomic dysreflexia and orthostatic hypotension | Baseline, prior to laboratory diagnostic testing session
  Participants will be given the Autonomic Dysfunction Following Spinal Cord Injury questionnaire (score range 0-436, with higher scores indicating more autonomic dysfunction).
Quantify secondary autonomic complications | Baseline, prior to laboratory diagnostic testing session
  Participants will be given the Composite Autonomic Symptom Score (range 0-100, with higher scores indicating more autonomic dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Solinsky, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No